CLINICAL TRIAL: NCT04598893
Title: A Multicenter, Multinational Extension of Study PRV-031-001 to Evaluate the Long-Term Safety of Teplizumab (PRV-031), a Humanized, FcR Non-Binding, Anti-CD3 Monoclonal Antibody, in Children and Adolescents With Recent-Onset Type 1 Diabetes Mellitus
Brief Title: Recent-Onset Type 1 Diabetes Extension Study Evaluating the Long-Term Safety of Teplizumab (PROTECT Extension)
Status: Active, not recruiting | Type: Observational
Sponsor: Provention Bio, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Other Study IDs: PRV-031-003
Record Dates: First submitted 2020-10-16; First posted 2020-10-22 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: Recent-onset type 1 diabetes; Teplizumab; T1D; Stage 3; Type 1 diabetes; New onset type 1 diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — teplizumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Teplizumab: Participants who received teplizumab in the PROTECT study
  Interventions: Biological: Teplizumab
- Placebo: Participants who received placebo in the PROTECT study
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Teplizumab — Received teplizumab in PROTECT Study
  Groups: Teplizumab
Other: Placebo — Received placebo in PROTECT study
  Groups: Placebo

SUMMARY:
The purpose of this non-interventional extension study is to continue to collect long-term safety and other clinical data for an additional 42 months in participants who completed the PROTECT study.

DETAILED DESCRIPTION:
This study is the long-term extension of the PRV-031-001 (PROTECT) study. PROTECT is a Phase 3, randomized, double-blind, placebo-controlled, multinational, multi-center study to evaluate the efficacy and safety of teplizumab, a humanized, anti-CD3 monoclonal antibody, in children and adolescents ages 8 through 17 recently diagnosed with type 1 diabetes (within 6 weeks of diagnosis) in which approximately 300 participants were randomized at a ratio of 2:1 to the teplizumab or placebo and received two courses of treatment administered 6 or 12 months apart with final follow-up at approximately 18 months (78 weeks) after the first dose.

Participants who complete the PROTECT study are invited to enroll in this observational, extension study to collect long-term safety and other clinical data. The decision to participate can be made within 12 months of completing the PROTECT study.

No study drug will be administered during this extension study. Participants will continue to receive standard care for type 1 diabetes from their primary physicians.

Participants will return to the study sites for assessments once every 6 months through Month 42. Therefore, the combined duration of the PROTECT and PROTECT Extension studies will be 60 months.

ELIGIBILITY:
Inclusion Criteria:

1. Completion of the PRV-031-001 (PROTECT) study by completing the Week 78 visit in that study, regardless of how many doses of study drug were administered.
2. Provide written informed consent within 12 months of the Week 78 in the PRV-031-001 study. Written assent will be obtained for participants under 18 years of age at the time of enrollment, according to applicable regulations. If possible, written informed consent and/or assent for the current PROTECT Extension study (PRV-031-003) should be obtained at the final (Week 78) visit in the PROTECT study.

Exclusion Criteria:

1. Premature discontinuation from the PRV-031-001 (PROTECT) study for any reason.

Ages: 9 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Participants who completed the PROTECT (PRV-031-001) study
Sampling Method: Non-Probability Sample
Enrollment: 188 (Actual)
Dates: Start 2020-10-26 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events (AEs), serious adverse events (SAEs) and adverse events of special interest (AESIs), including infections and malignancies | During 42 months of follow-up
  Safety outcome

SECONDARY OUTCOMES:
Area under the time-versus concentration curve (AUC) of C-peptide after a 4-hour (4h) mixed-meal tolerance test (MMTT) | During the 42 months of follow-up
  Clinical parameters of diabetes management 1
Insulin use (daily average insulin dose in U/kg/day) | During the 42 months of follow-up
  Clinical parameters of diabetes management 2
HbA1c | During the 42 months of follow-up
  Clinical parameters of diabetes management 3

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (47):
- United States (25):
  - Rady Children's Hospital 3020 Children's Way (Site 840004), San Diego, California
  - UCSF Medical Center Gateway Medical Building, 1825 Fourth Street (Site 840001), San Francisco, California
  - Diablo Clinical Research2255 Ygnacio Valley Road, Ste. M (Site 840002), Walnut Creek, California
  - Barbara Davis Center for Diabetes - Pediatrics 1775 Aurora Court (Site 840005), Aurora, Colorado
  - Nemours Children's Health, 807 Children's Way, Jacksonville, Florida
  - Johns Hopkins All Children's Hospital, 501 6th Avenue South (Site 840048), St. Petersburg, Florida
  - Atlanta Diabetes Associates 1800 Howell Mill Road. Suite 450 (Site 840009), Atlanta, Georgia
  - Centricity Research (Site 840006), Columbus, Georgia
  - St. Luke's Children's Endocrinology, 305 E Jefferson St. (Site 840052), Boise, Idaho
  - Rocky Mountain Clinical Research, LLC 3910 Washington Parkway, Suite E (Site 840007), Idaho Falls, Idaho
  - Indiana University Hospital, Indiana Clinical Research Center, 550 North University Boulevard (Site 840014), Indianapolis, Indiana
  - University of Iowa Hospitals and Clinics 200 Hawkins Drive (Site 840023), Iowa City, Iowa
  - Capital Medical Research Associates (Site 840029), Camp Springs, Maryland
  - Baystate Medical Center, 759 Chestnut Street, Springfield, Massachusetts
  - Children's Mercy Hospitals and Clinics, 2401 Gillham Road (Site 840026), Kansas City, Missouri
  - Washington University School of Medicine, Pediatric Clinical Research Unit, Suite 11W19 (Site 840018), St Louis, Missouri
  - UBMD Pediatrics 1001 Main Street, 4th Floor (Site 840010), Buffalo, New York
  - UNC Hospitals, The University of North Carolina at Chapel Hill, Children's Specialty Clinic, 101 Manning Drive (Site 840038), Chapel Hill, North Carolina
  - Endocrinology Service Northwest, LLC 929 SW Simpson Ave. Suite 220 (Site 840034), Bend, Oregon
  - Children's Hospital of Philadelphia, Division of Endocrinology 3500 Civic Center Blvd., Buerger Center 12th Floor (Site 840021), Philadelphia, Pennsylvania
  - AM Diabetes & Endocrinology Center, 3025 Kate Bond Rd. (Site 840008), Bartlett, Tennessee
  - Vanderbilt University Medical Center 1500 21st Avenue, Suite 1514, Village At Vanderbilt (Site 840024), Nashville, Tennessee
  - UT Southwestern Children's Medical Center of Dallas 1935 Medical District Drive (Site 840033), Dallas, Texas
  - Virginia Mason Medical Center, Benaroya Research Institute 1201 9th Ave, MS: D4-CRP (Site 840016), Seattle, Washington
  - MultiCare Health System, Gateway Medical Building (Site 840003), Tacoma, Washington
- Belgium (2):
  - University Hospital Brussels (Site 056202), Jette, Brussels Capital
  - UCL Namur University Hospital Place Louise Godin 15 (Site 056205), Namur, Namur
- Canada (2):
  - Alberta Diabetes Institute, 2-004 Li Ka Shing Centre for Health Research Innovation 8602 (Site 124103), Edmundston, Alberta
  - BCDiabetes - Medical Research Center, 210 West Broadway Suite 400 (Site 124102), Vancouver, British Columbia
- University Hospital Motol V Uvalu 84, Praha 5 - Motol (Site 203301), Prague, Czechia
- France (7):
  - Hospital Center Regional D'Orleans Hospital La Source, Pediatric Department, 14 Hospital Ave Post box 86709 (Site 250513), Orléans, France
  - Woman Mother Child Hospital HCL, Bron
  - Dijon University Hospital Center-Francois Mitterand Hospital, Children's Hospital, Dijon
  - CHU La Timone - La Timone Children's Hospital, Marseille
  - Lenval Hospital, 57 Avenue de la Californie (Site 250508), Nice
  - Necker Children's Hospital, 149 Rue de Sevres (Site 250502), Paris
  - Pau Hospital Center, Pau
- Germany (5):
  - Evangelic Clinic Bethel, Children's Clinic Grenzweg 14/Hs 2 (Site 276602), Bethel, Bielefeld
  - Hospital Augsburg, Stenglinstrasse 2 (Site 276606), Augsburg
  - University Hospital Carl Gustav Carus Fetscherstrasse 74 (Site 276601), Dresden
  - Pediatric Hospital on the Bult Janusz-Korczak-Allee 12 (Site 276604), Hanover
  - University Hospital Heidelberg, Im Neuenheimer Feld 430 (Site 276608), Heidelberg
- Poland (4):
  - University Teaching Centre of the Medical University of Warsaw, 63A, ul. Zwirki i Wigur (Site 616804), Warsaw, Poland
  - University Teaching Centre, Department of Pediatrics, Diabetology and Endocrinology (Site 616803), Gdansk
  - Institute of Diabetology ul. Raclawicka 129/2U, 02-117 (Site 616802), Warsaw
  - Children's Memorial Health Institute Al. Dzieci Polskich 20 (Site 616801), Warsaw
- Sheffield Children's Hospital Western Bank, S10 2TH (Site 826903), Sheffield, Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org